CLINICAL TRIAL: NCT06792513
Title: The Effectiveness of Acrylic and Clear Aligners in the Treatment of Anterior Crossbite in Children And Evaluatıon of The Effects of These Treatments on Quality of Life
Brief Title: The Effectiveness of Acrylic and Clear Aligners in the Treatment of Anterior Crossbite in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ozge Gungor (Other)
Collaborators: Akdeniz University (Other)
Responsible Party: Sponsor-Investigator, Ozge Gungor, PhD, DDS, Clinical Associate Professor of Pedodontics, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUBNG001
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Anterior Crossbite
Keywords: anterior crossbite; cephalometric analysis; clear aligners; labiolingual spring Hawley; quality of life
MeSH Terms: interventions — Orthodontic Appliances, Removable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clear aligner (group treated with clear aligner) (Experimental): 2 parallel groups one treated with clear aligner and other treated using labiolingual spring Hawley appliances
  Interventions: Device: Clear Aligner
- Labiolingual spring Hawley appliances (group treated with labiolingual spring Hawley appliances) (Experimental): 2 parallel groups one treated with clear aligner and other treated using labiolingual spring Hawley appliances
  Interventions: Device: Labiolingual Spring Hawley Appliance

INTERVENTIONS:
Device: Clear Aligner — In this intervention, clear aligners were digitally designed using three-dimensional models for the upper jaw. Attachments were applied to the patients, specifically placed on the incisors exhibiting a crossbite relationship and on the permanent first molars in the posterior region. The series of clear aligners were replaced every 10 days. The aligners were used full-time, except during meals and tooth brushing.
  Arms: Clear aligner (group treated with clear aligner)
Device: Labiolingual Spring Hawley Appliance — In this intervention, a custom-made labiolingual spring Hawley appliance was designed for the upper jaw. It included two Adams clasps, a vestibular arch, and an active labiolingual spring positioned on the palatal side of the incisor in crossbite. The spring was activated every 10 days. The appliance was used full-time, except during meals and tooth brushing.
  Other Names: Z spring appliance
  Arms: Labiolingual spring Hawley appliances (group treated with labiolingual spring Hawley appliances)

SUMMARY:
To evaluate the treatment efficacy, treatment duration, and cephalometric changes, as well as the impact on quality of life, of clear aligners and labiolingual spring Hawley appliances in the treatment of pediatric patients with anterior crossbite.

DETAILED DESCRIPTION:
Two groups were treated with clear aligners and labiolingual springs Hawley and the study consisted of 30 patients, 15 patients in each group. Cast analysis and cephalometric analysis were performed at pretreatment and posttreatment. Quality of life was assessed at the end of treatment for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. In the mixed dentition phase, aged between 7-12 years
2. With a dental Class I molar relationship according to Angle's classification
3. ANB within the normal range i.e. (the crossbite will be diagnosed as dental)
4. Exhibiting anterior crossbite (AC) in at least one permanent incisor in the sagittal plane
5. No prior orthodontic treatment for any reason
6. No history of maxillofacial trauma
7. No systemic diseases or syndromes that may interfere with treatment
8. Able to attend regular appointments and cooperate with instructions throughout the treatment process

Exclusion Criteria:

1. Patients with functional anterior crossbite associated with mandibular functional shift
2. Patients with clinically evident retrognathia or prognathia of the maxilla or mandible
3. Patients with severe gingivitis or periodontitis
4. Patients with known allergies to the materials to be used in the treatment
5. Patients with severe dental anomalies (e.g., supernumerary teeth, missing teeth, dental malformations)
6. Patients with serious emotional or psychological issues that may hinder treatment compliance

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Changes in Cephalometric Measurements Before and After Treatment Assessed Using Dolphin Imaging Software (Version 11.95) | 3 months
  Comparison of cephalometric measurements (e.g., ANB, FMA, U1-NA angle, overjet, and overbite) between the two groups at pre-treatment and post-treatment periods. Measurements will be performed using Dolphin Imaging Software version 11.95, with units reported in degrees and millimeters as applicable.
Changes in Oral Health-Related Quality of Life Assessed Using the Child Oral Health Impact Profile-Short Form 19 (COHIP-SF-19) | 3 months
  COHIP-SF-19 scores will be assessed at the end of the treatment period to evaluate changes in oral health-related quality of life. The scale ranges from 0 to 76, with higher scores indicating worse oral health-related quality of life.

SECONDARY OUTCOMES:
Changes in Analogue Cast Model Measurements Before and After Treatment | 3 months
  Comparison of analogue model measurements, including parameters such as arch depth and arch length, between the two groups at pre-treatment and post-treatment periods. Measurements will be performed using calipers on analogue cast models. Units of measure include millimeters (mm).
3D model measurements | 3 months
  Comparison of the measurements of the 3D digital model analysis of the two groups at the pre-treatment and at the post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Özge Güngör, PhD, DDS, Assoc. Prof., Study Director — Akdeniz University Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Akdeniz University Faculty of Dentistry, Department of Pediatric Dentistry, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
A final decision regarding the sharing of individual participant data (IPD) has not yet been made. Appropriate data-sharing protocols will be evaluated in the future before reaching a decision.